CLINICAL TRIAL: NCT04443270
Title: Efficacy of Chloroquine Phosphate Prophylactic Use in First-line Health Personnel Exposed to COVID-19 Patients
Brief Title: Chloroquine Phosphate Prophylactic Use in Health Personnel Exposed to COVID-19 Patients
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: CMN "20 de Noviembre" (Other)
Responsible Party: Principal Investigator, Sandra Muñoz López, Internal Medicine Service Member, MD, MSc, CMN "20 de Noviembre"
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 01
Record Dates: First submitted 2020-06-17; First posted 2020-06-23 (Actual); Last update posted 2020-07-14 (Actual); Status verified 2020-07

CONDITIONS: COVID-19
Keywords: COVID-19; Chloroquine phosphate; Prophylactic; Health Personnel; Severe Acute Respiratory Syndrome Coronavirus-2
MeSH Terms: conditions — COVID-19 | interventions — chloroquine diphosphate

STUDY DESIGN:
Intervention Model Description: Controlled Clinical Trial
Who Masked: Outcomes Assessor
Masking Description: The Outcome Assessor will be an external member of the Internal Medicine Service, which will be blinded to the intervention.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Chloroquine phosphate prophylactic group (Experimental): Drug: Chloroquine phosphate
  Dosage form, frequency and duration: 300 mg per day during initial 30 days and 150 mg per day during the next 30 days.
  Interventions: Drug: Chloroquine phosphate
- Control group (No Intervention): Health personnel who want to be included voluntary in the study and meet the inclusion criteria without Chloroquine use.

INTERVENTIONS:
Drug: Chloroquine phosphate — Drug: Chloroquine phosphate
  Dosage form, frequency and duration: 300 mg per day during initial 30 days and 150 mg per day during the next 30 days.
  Other Names: Plasmodín
  Arms: Chloroquine phosphate prophylactic group

SUMMARY:
The primary objective of this study is to evaluate the efficacy and security of chloroquine phosphate prophylactic use for reducing the risk of infection by severe acute respiratory syndrome coronavirus-2 in Health Care Workers exposed to COVID-19 patients.

DETAILED DESCRIPTION:
Health Care Workers as first line of hospital care, are at high risk of infection by severe acute respiratory syndrome coronavirus-2 due for the exposure to COVID-19 patients. The pharmacological treatment with chloroquine phosphate has emerged as one of the main therapeutic approaches for COVID-19 patients. However, some studies have described and hypothesized that the use of prophylactic chloroquine phosphate could provide some protection against COVID-19 infection reducing the chances of contagion in Health Care personnel during the development of the pandemic. A controlled clinical trial will be conducted in a tertiary hospital in Mexico City, Mexico. Participants will be divide in two groups; 1) intervention: who will receive chloroquine phosphate (300 mg/day during the first 30 days and 150mg/day during the last 30 days) and 2) control, both with a follow up for 60 days.

ELIGIBILITY:
Inclusion Criteria:

* Health Care Workers as first line of hospital care exposed to COVID-19 patients.
* Initial polymerase chain reaction assay negative test for severe acute respiratory syndrome coronavirus-2 infection.
* Both sexes
* Agree to participate in the study after signing an informed consent letter.

Exclusion Criteria:

* Health Care Workers as first line of hospital care exposed to COVID-19 patients with history of heart disease, arrhythmias or QT segment prolongation.
* Health Care Workers as first line of hospital care exposed to COVID-19 patients with liver or kidney disease of any etiology.
* Health Care Workers as first line of hospital care exposed to COVID-19 patients with retinopathy of any etiology.
* Health Care Workers as first line of hospital care exposed to COVID-19 patients with allergy to chloroquine.
* Health Care Workers as first line of hospital care exposed to COVID-19 patients with a history or diagnosis of psoriasis.
* Health Care Workers as first line of hospital care exposed to COVID-19 patients with important primary clinical alterations: renal (creatinine> 3), liver (Alanine Aminotransferase and Aspartate Aminotransferase x 3), endocrine, neurological.

Ages: 18 Years to 59 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 200 (Estimated)
Dates: Start 2020-07-27 (Estimated); Primary Completion 2020-10-31 (Estimated); Study Completion 2021-01-31 (Estimated)

PRIMARY OUTCOMES:
Negative Polymerase Chain Reaction assay at day 0 | Day 0
  Prior to the participation of each health worker, a pharyngeal exudate sample will be taken with a swab. RNA will be obtained by applying severe acute respiratory syndrome coronavirus-2 real time polymerase chain reaction kit, using specific oligonucleotides in polymerase chain reaction.
Polymerase Chain Reaction assay at day 60 | Day 60
  A pharyngeal exudate sample will be taken with a swab. RNA will be obtained by applying severe acute respiratory syndrome coronavirus-2 real time polymerase chain reaction kit, using specific oligonucleotides in polymerase chain reaction.

SECONDARY OUTCOMES:
Clinical improvement related to COVID-19 | Baseline (day 0) and 30-day follow up
  Ordinal Scale for Clinical Improvement according the "World Health Organization R&D Blueprint novel Coronavirus COVID-19 Therapeutic Trial Synopsis" will apply at baseline and 30-day follow-up as follows:
  No clinical or virological evidence of infection = 0 No limitation of activities = 1 Limitation of activities = 2 Hospitalized, no oxygen therapy = 3 Oxygen by mask or nasal prongs = 4 Non-invasive ventilation or high-flow oxygen = 5 Intubation and mechanical ventilation - Score = 6 Ventilation + additional organ support-pressors, renal replacement therapy, extracorporeal membrane oxygenation = 7 Death = 8
Clinical improvement related to COVID-19 | From 30-day to 60-day follow-up
  Ordinal Scale for Clinical Improvement according the "World Health Organization R&D Blueprint novel Coronavirus COVID-19 Therapeutic Trial Synopsis" will apply at baseline and 30-day follow-up as follows:
  No clinical or virological evidence of infection = 0 No limitation of activities = 1 Limitation of activities = 2 Hospitalized, no oxygen therapy = 3 Oxygen by mask or nasal prongs = 4 Non-invasive ventilation or high-flow oxygen = 5 Intubation and mechanical ventilation - Score = 6 Ventilation + additional organ support-pressors, renal replacement therapy, extracorporeal membrane oxygenation = 7 Death = 88
Heart rhythm negative adverse event related to the Chloroquine Phosphate Prophylactic Use | Baseline (day 0) and 30-day follow up
  An EKG will be performed to measure QT interval at baseline and 30-day follow-up.
  The EKG follows the standards and guidelines established by the Centro Médico Nacional "20 de Noviembre."
Heart rhythm negative adverse event related to the Chloroquine Phosphate Prophylactic | From 30-day to 60-day follow-up
  An EKG will be performed to measure QT interval at 60-day follow-up.
  The EKG follows the standards and guidelines established by the Centro Médico Nacional "20 de Noviembre."
COVID-19 symptomatic onset rate | From baseline (day 0) to 60-day follow up
  According to the National Committee for Epidemiological Surveillance (CONAVE) in Mexico, COVID-19 symptomatic onset rate defined as the presence of cough, fever or headache during the last 7 days, accompanied at least one of the following symptoms: dyspnea, arthralgia, myalgia, odynophagia / pharyngeal burning, rhinorrhea, conjunctivitis or chest pain.

CONTACTS AND LOCATIONS:
Overall Officials: Sandra Muñoz-López, MD, MSc, Principal Investigator — CMN "20 de Noviembre"; Sandra Muñoz-López, MD, MSc, Study Director — CMN "20 de Noviembre"; Maricela Escarela-Serrano, MD, Study Chair — CMN "20 de Noviembre"; Fedra Irazoque-Palazuelos, MD, Study Chair — CMN "20 de Noviembre"; Luis Montiel-López, MD, MSc, Study Chair — CMN "20 de Noviembre"; Paul Mondragón-Terán, PhD, Study Chair — CMN "20 de Noviembre"; Alberto H De la Vega-Bravo, MD, Study Chair — CMN "20 de Noviembre"; Juan A Pineda-Juárez, PhD, Study Chair — CMN "20 de Noviembre"; Juan A Suárez-Cuenca, MD, PhD, Study Chair — CMN "20 de Noviembre"; Sofía L Alcaraz-Estrada, PhD, Study Chair — CMN "20 de Noviembre"; Eduardo Soei-Sarmiento, BsC, Study Chair — CMN "20 de Noviembre"; Maribel Santosbeña-Lagunes, MD, Study Chair — CMN "20 de Noviembre"; Joel Vargas-Hernández, MD, Study Chair — CMN "20 de Noviembre"; Carlos A Delgado-Quintana, MD, Study Chair — CMN "20 de Noviembre"; Alejandro Alanis-Vega, MD, Study Chair — CMN "20 de Noviembre"; Ricardo P Vázquez-Alvarado, MD, Study Chair — CMN "20 de Noviembre"; Mireya Rodríguez-Martínez, MD, Study Chair — CMN "20 de Noviembre"; María C Méndez-Vidrio, MD, Study Chair — CMN "20 de Noviembre"; Fidel Cerda-Tellez, MD, Study Chair — CMN "20 de Noviembre"
Locations (1):
- Centro Médico Nacional "20 de Noviembre", Mexico City, Benito Juárez, Mexico

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Rothan HA, Byrareddy SN. The epidemiology and pathogenesis of coronavirus disease (COVID-19) outbreak. J Autoimmun. 2020 May;109:102433. doi: 10.1016/j.jaut.2020.102433. Epub 2020 Feb 26. PMID 32113704
- [Background] Adhikari SP, Meng S, Wu YJ, Mao YP, Ye RX, Wang QZ, Sun C, Sylvia S, Rozelle S, Raat H, Zhou H. Epidemiology, causes, clinical manifestation and diagnosis, prevention and control of coronavirus disease (COVID-19) during the early outbreak period: a scoping review. Infect Dis Poverty. 2020 Mar 17;9(1):29. doi: 10.1186/s40249-020-00646-x. PMID 32183901
- [Background] Singhal T. A Review of Coronavirus Disease-2019 (COVID-19). Indian J Pediatr. 2020 Apr;87(4):281-286. doi: 10.1007/s12098-020-03263-6. Epub 2020 Mar 13. PMID 32166607
- [Background] Sohrabi C, Alsafi Z, O'Neill N, Khan M, Kerwan A, Al-Jabir A, Iosifidis C, Agha R. World Health Organization declares global emergency: A review of the 2019 novel coronavirus (COVID-19). Int J Surg. 2020 Apr;76:71-76. doi: 10.1016/j.ijsu.2020.02.034. Epub 2020 Feb 26. PMID 32112977
- [Background] Kannan S, Shaik Syed Ali P, Sheeza A, Hemalatha K. COVID-19 (Novel Coronavirus 2019) - recent trends. Eur Rev Med Pharmacol Sci. 2020 Feb;24(4):2006-2011. doi: 10.26355/eurrev_202002_20378. PMID 32141569
- [Background] Lai CC, Shih TP, Ko WC, Tang HJ, Hsueh PR. Severe acute respiratory syndrome coronavirus 2 (SARS-CoV-2) and coronavirus disease-2019 (COVID-19): The epidemic and the challenges. Int J Antimicrob Agents. 2020 Mar;55(3):105924. doi: 10.1016/j.ijantimicag.2020.105924. Epub 2020 Feb 17. PMID 32081636
- [Background] Ahn DG, Shin HJ, Kim MH, Lee S, Kim HS, Myoung J, Kim BT, Kim SJ. Current Status of Epidemiology, Diagnosis, Therapeutics, and Vaccines for Novel Coronavirus Disease 2019 (COVID-19). J Microbiol Biotechnol. 2020 Mar 28;30(3):313-324. doi: 10.4014/jmb.2003.03011. PMID 32238757
- [Background] Gao J, Tian Z, Yang X. Breakthrough: Chloroquine phosphate has shown apparent efficacy in treatment of COVID-19 associated pneumonia in clinical studies. Biosci Trends. 2020 Mar 16;14(1):72-73. doi: 10.5582/bst.2020.01047. Epub 2020 Feb 19. PMID 32074550
- [Background] Gautret P, Lagier JC, Parola P, Hoang VT, Meddeb L, Mailhe M, Doudier B, Courjon J, Giordanengo V, Vieira VE, Tissot Dupont H, Honore S, Colson P, Chabriere E, La Scola B, Rolain JM, Brouqui P, Raoult D. RETRACTED: Hydroxychloroquine and azithromycin as a treatment of COVID-19: results of an open-label non-randomized clinical trial. Int J Antimicrob Agents. 2020 Jul;56(1):105949. doi: 10.1016/j.ijantimicag.2020.105949. Epub 2020 Mar 20. PMID 32205204
- [Background] Principi N, Esposito S. Chloroquine or hydroxychloroquine for prophylaxis of COVID-19. Lancet Infect Dis. 2020 Oct;20(10):1118. doi: 10.1016/S1473-3099(20)30296-6. Epub 2020 Apr 17. No abstract available. PMID 32311322
- [Background] Rathi S, Ish P, Kalantri A, Kalantri S. Hydroxychloroquine prophylaxis for COVID-19 contacts in India. Lancet Infect Dis. 2020 Oct;20(10):1118-1119. doi: 10.1016/S1473-3099(20)30313-3. Epub 2020 Apr 17. No abstract available. PMID 32311324
- [Background] Gendrot M, Javelle E, Clerc A, Savini H, Pradines B. Chloroquine as a prophylactic agent against COVID-19? Int J Antimicrob Agents. 2020 Jun;55(6):105980. doi: 10.1016/j.ijantimicag.2020.105980. Epub 2020 Apr 12. PMID 32294495
- See also: World Health Organization. Coronavirus disease (COVID-19) outbreak situation. — https://www.who.int/emergencies/diseases/novel-coronavirus-2019
- See also: World Health Organization. Rolling updates on coronavirus disease (COVID-19). — https://www.who.int/emergencies/diseases/novel-coronavirus-2019/events-as-they-happen
- See also: FDA cautions against use of hydroxychloroquine or chloroquine for COVID-19 outside of the hospital setting or a clinical trial due to risk of heart rhythm problems. 2020. — https://www.fda.gov/drugs/drug-safety-and-availability/fda-cautions-against-use-hydroxychloroquine-or-chloroquine-covid-19-outside-hospital-setting-or